CLINICAL TRIAL: NCT02569138
Title: Investigating Long Term Balance-Enhancing Effects of Insole Hardness and Thickness for Older Adult Footwear
Brief Title: Balance-Enhancing Effects of Insole Hardness and Thickness for Older Adult Footwear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Dr. Stephen Perry, Professor, Wilfrid Laurier University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EM_FFP
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Accidental Falls
Keywords: Balance; Footwear; Shoes; Falls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insole (Experimental) (Experimental): specially designed insole, featuring hard and thin design, modified insole
  Interventions: Device: Modified Insole
- Insole (Control) (Experimental): usual insole found in footwear, non-modified insole
  Interventions: Device: Non-Modified Insole

INTERVENTIONS:
Device: Modified Insole — hard and thin shoe insert between the foot sole and base of the footwear
  Arms: Insole (Experimental)
Device: Non-Modified Insole — regular shoe insert between the foot sole and base of the footwear
  Arms: Insole (Control)

SUMMARY:
The purpose of this study is to investigate the long term balance-enhancing effects of insoles that are hard and thin for older adults. Thirty older female adults between the ages of 65-84 years will be recruited for this study. Twenty participants (20) will wear the experimental insole and ten (10) participants will work their usual insole, during a 12 week period. Balance and foot sensitivity testing will take place at 0, 6 and 12 weeks. These tests will involve measurement of body motion and foot pressure in order to evaluate balance control. Additionally, each participant will be asked to return a bi-weekly postcard that will report on footwear wearing patterns and any falls (or fall-related) incidents that have occurred during the 12 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the long term balance-enhancing effects of insoles that are hard and thin for older adults. Thirty older female adults between the ages of 65-84 years will be recruited for this study. Those who are defined as healthy older adults as per the initial screening questionnaire will be asked to complete additional screening tests during a scheduled testing session including sensory testing, balance testing, and cognitive testing using monofilaments, the Berg Balance Scale, and the Montreal Cognitive Assessment tool, respectively. Participants will also be examined for degree of hallux valgus using the Manchester Scale, since moderate to severe hallux valgus has displayed balance deficits for older adults. Those participants that complete all tests and display acceptable age range scores as define by the test guidelines will be randomly selected to either be in an intervention group (20 participants) or a control group (10 participants). All participants will be fitted for custom insoles that are hard and thin. These insoles will not affect their habitual ankle position or habitual stance in any way. These insoles will be designed to mechanically support the foot within the shoe, but mostly to provide as much somatosensory feedback as possible detected through mechanoreceptors under the skin on the plantar sole of the foot. Participants in the intervention group will be required to wear these insoles in their shoes for the full 12 week intervention. One pair of each participant's shoes of both groups will be chosen by the primary investigator to be worn for the entire duration of the 12 week intervention for at least 8 hours per day. These shoes will be chosen if eligible within a footwear assessment form and previous footwear recommendations from previous literature for older adults. Each testing session will be held in a common room located within close vicinity of the participant's residence. A camcorder will be used to record participant movement during each trial located directly in front of the participant. Foam markers will then be fastened on to the participant's body using tape at 7 locations to allow for body movement analysis in correspondence with the video recording. Flat and thin pressure sensor insoles that will not cause any discomfort to the participant will be place into each shoe to detect the pressure forces and distribution under the feet. Once equipment has been set up in the room and with the participant, participants will complete various tasks including quiet standing, one-legged stance, and walking up and down a ramp while unexpectedly terminating gait (10 seconds), performing a cognitive task while walking up and down a ramp (10 seconds), and normal walking (10 seconds). Participants will be provided with 12 postcards outlining general questions regarding insole and footwear comfort, hours of wear, and record of falls. Participants will be required to complete these cards twice a week and mail/return the cards to Wilfrid Laurier University. The cards will be pre-printed with address on the front and a sticky tab to seal the card once completed.

ELIGIBILITY:
Inclusion Criteria:

* have appropriate footwear

Exclusion Criteria:

* any vestibular, neurological, or muscular injuries that may affect their balance or gait

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change of Stability Margin from Week 0 | At 0, 6, and 12 Weeks
  Stability margin is the ability of the individual to maintain their body's balance point within their base of support while walking or performing a balance task

SECONDARY OUTCOMES:
Number of Falls | Recorded twice a week during the 12 week study duration

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McLeod, BSc, Principal Investigator — Wilfrid Laurier University
Locations (1):
- Biomechanics Lab, Wilfrid Laurier University, Waterloo, Ontario, Canada